CLINICAL TRIAL: NCT06473753
Title: Clinical and Neurophysiological Assessment of Pelvic Floor Dysfunction in Patients With Multiple Sclerosis
Brief Title: Pelvic Floor Disorders in Multiple Sclerosis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yosra Abdallah Hassan, Principal investigator, Assiut University
Other Study IDs: M.s pelvic floor disorders
Record Dates: First submitted 2023-12-06; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Primary objective

1. Clinical assessment of bowel, bladder, and sexual dysfunction in patients with MS
2. Impact of sphincter disorders on quality of life in patients with MS by using correlation between Extended Disability Status Scale (EDSS)and The Incontinence Quality of Life Questionnaire (IQOL)

Secondary objectives

-Studying the effect of low frequency rTMS on bladder symptoms in patients with MS.

DETAILED DESCRIPTION:
2.4.1- Type of the study: This study will be a cross-section observational study. 2.4. 2- Study Setting: neuology unit assuit university hospital 2.4. 3- Study subjects: From the neurologic outpatient clinic in Assiut University and patients referred from our staff members in Neuropsychiatry department.

1. Inclusion criteria:

   Adult patient with definite Multiple sclerosis according to Mcdonald's Criteria (revised criteria 2017), Age > 18 years both sexes patient with subjective complaint of any of pelvic floor dysfunction (bladder, sexual or bowel)
2. Exclusion criteria:

Patients with other systemic or neurological disorder affecting sphincter (Diabetes Mellitus, Renal diseases, Urinary tract infection, epilepsy, peripheral neuropathy, irritable bowel syndrome…..) Patients taking drugs affecting sphincter as psychotropic drugs

2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): Step I Patients will be assessed through full neurological history and examination with

All of them will be subjected to the following scales:

* Extended Disability Status Scale (EDSS)
* Multiple Sclerosis Quality of Life Inventory (MSQLI)
* Actionable Bladder Symptom Screening Tool (ABSST)
* Neurogenic Bladder Symptom Score (NBSS)
* The Incontinence Quality of Life Questionnaire (IQOL)
* Neurogenic Bowel Dysfunction Score (NBD)
* Multiple sclerosis intimacy and sexuality questionnaire 19-item version (MSISQ-19) Step II All patients will have the paraclinical assessment in form of neuroimaging (recent MRI brain and spine within last year) evoked potentials (visual, auditory brainstem) Motor evoked potential using TMS with parameters gained using single pulse paradigm Step III as a fulfillment for our secondary objective regarding the study of the effect of rTMS on urinary dysfunction we will recruit 20 patients with significant urinary dysfunction according to assessment results with EDSS ≤ 6 and they will be randomized in two arms for active and sham application of rTMS. by using high intensity low frequency protocol for rTMS application[39] for 10 sessions over two weeks with using voiding diary, specific selected scales and selected cortical excitability measures as assessment tools, we will follow up the patients immediately and for one month post sessions.

ELIGIBILITY:
Inclusion Criteria:

1.Adult patient with definite Multiple sclerosis 2-Age > 18 years 3-both sexes 4-patient with complaint of any of pelvic floor dysfunction (bladder, sexual or bowel)

Exclusion Criteria:

1. Patients with other systemic or neurological disorder affecting sphincter.
2. Patients taking drugs affecting sphincter.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with multiple sclerosis according to McDonald's criteria 2017 attending outpatient clinic, department of neurology and psychiatry, Assuit university hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of bowel, bladder, and sexual dysfunction in patients with MS though applying specific related scales | Baseline
  Clinical assessment of bowel, bladder, and sexual dysfunction in patients with MS though applying specific related scales

SECONDARY OUTCOMES:
Motor evoked potential using TMS with parameters gained using single pulse paradigm | Baseline
  Motor evoked potential using TMS with parameters gained using single pulse paradigm effect on sphincter distrubance in multiple sclerosis.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Belbasis L, Bellou V, Evangelou E, Tzoulaki I. Environmental factors and risk of multiple sclerosis: Findings from meta-analyses and Mendelian randomization studies. Mult Scler. 2020 Apr;26(4):397-404. doi: 10.1177/1352458519872664. Epub 2019 Sep 6. PMID 32249718